CLINICAL TRIAL: NCT02367924
Title: Non-interventional Study to Investigate Efficacy and Safety of Trabectedin (Yondelis®) in Patients With Advanced Soft Tissue Sarcoma
Brief Title: Efficacy and Safety of Trabectedin (Yondelis®) in Patients With Advanced Soft Tissue Sarcoma
Acronym: YonSar
Status: Completed | Type: Observational
Sponsor: PharmaMar, Spain (Industry)
Responsible Party: Sponsor
Other Study IDs: ET-D-023-13
Record Dates: First submitted 2015-02-04; First posted 2015-02-20 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Yondelis: The administration of chemotherapy regimen with trabectedin (according to Summary of Product Characteristics (SmPC)) will be determined by the Investigator's discretion depending on the patients' conditions and previous chemotherapy.
  Interventions: Drug: trabectedin

INTERVENTIONS:
Drug: trabectedin — The administration of chemotherapy regimen with trabectedin (according to Summary of Product Characteristics (SmPC)) will be determined by the Investigator's discretion depending on the patients' conditions and previous chemotherapy.
  Other Names: Yondelis

SUMMARY:
Efficacy and safety of trabectedin in real-life practice, routinely used for the management of advanced sarcoma after failure of anthracyclines and ifosfamide or patients unsuited to receive these drugs in Germany.

Trabectedin is indicated for the treatment of patients with advanced soft tissue sarcoma, after failure of anthracyclines and ifosfamide, or who are unsuited to receive these agents. Efficacy data are based mainly on liposarcoma and leiomyosarcoma patients.

DETAILED DESCRIPTION:
This is a non-interventional, observational and prospective study to evaluate efficacy and safety of trabectedin in routine practice. Patients are assigned to a therapeutic strategy within current practice, not according to a trial protocol. The prescription of the medicine is separated from the decision to include the patient in the study. Diagnostic or monitoring procedures are only those ordinarily applied to the therapeutic strategy.

There are no dose regimens or medical procedures defined within this study plan. Every medical decision and course of treatment with trabectedin will reflect exclusively the decision of the Investigator in a routine clinical situation according to SmPC. The concept of this non-interventional study and its documentation procedure will not affect in any way the routine treatment situation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must comply with all of the following criteria in order to be enrolled into the study:

  * Histologically diagnosed advanced STS
  * Female or male aged 18 years or above
  * Signed written informed consent
  * Suitable to undergo treatment with trabectedin according to SmPC
  * Progress after therapy with anthracyclines and ifosfamide has failed, or if patients are unsuited to receive these agents

Exclusion Criteria:

* Patients presenting contraindications for the use of trabectedin as defined in the SmPC will be excluded from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients (≥ 18 years) with advanced sarcoma after failure of anthracyclines and ifosfamide or patients unsuited to receive these drugs
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
3 months progression free survival (PFS) rate | 3 months after start of therapy
  Number of patients without PD or death 3 months after start of therapy
6 months progression free survival (PFS) rate | 6 months after start of therapy
  Number of patients without PD or death 6 months after start of therapy

SECONDARY OUTCOMES:
Tumor control rate | in average 6 months
  Best response (CR+PR+Disease stabilization) according to institutional standards
3 and 6 months overall survival (OS) rate | 3 and 6 months after start of therapy
  Number of patients alive after 3 months and 6 months
Progression free survival (PFS) | in average 6 months
  Time from start of therapy to the date of documented PD or death (death of any cause)
Type of treatment used | 2 years
  dose reductions and postponement of cycles
Treatment duration | from first cycle up to a maximum of 17 cycles, each cycle is 21 days (= 1 year)
  Number of cycles
Reason for discontinuation of trabectedin treatment | from first cycle up to a maximum of 17 cycles, each cycle is 21 days (= 1 year)
  Analysis of documented reasons
General description of grade 3/4 adverse events | 2 years
  Adverse events of grade 3/4 according to NCI CTC V4

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Grünwald, Dr., Principal Investigator — Hannover Medical School
Locations (19):
- Germany (19):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinikum der Landeshauptstadt Stuttgart gKAöR - Klinik für Onkologie, Stuttgart, Baden-Wurttemberg
  - Universitätsklinikum Augsburg A.d.ö.R - II. Medizinische Klinik, Augsburg, Bavaria
  - Onkologisches Zentrum Donauwörth, Donauwörth, Bavaria
  - LMU - Klinikum der Universität München - Medizinische Klinik und Poliklinik III/Hämatologie und Onkologie, München, Bavaria
  - Klinikum Nürnberg Nord - Medizinische Klinik 5, Schwerpunkt Onkologie/Hämatologie, Nuremberg, Bavaria
  - Universitätsklinikum Würzburg - Medizinische Klinik und Poliklinik II, Würzburg, Bavaria
  - HELIOS Klinikum Bad Saarow, Bad Saarow, Brandenburg
  - Lahn-Dill-Kliniken GmbH, Wetzlar, Hesse
  - Medizinische Hochschule Hannover - Klinik für Hämatologie, Hämostaseologie, Onkologie und Stammzelltransplantation, Hanover, Lower Saxony
  - Gemeinschaftspraxis Dr. Reichert, Dr. Janssen, Westerstede, Lower Saxony
  - Praxis Dr. Rodemer, Wilhelmshaven, Lower Saxony
  - MVZ Marien-Hospital-Wesel GmbH, Wesel, North Rhine-Westphalia
  - Universitätsklinikum Magdeburg A.ö.R., Magdeburg, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Charité - Universitätsmedizin Berlin, Berlin
  - Praxis für Innere Medizin, Hämatologie u. Onkologie, Bremen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Onko-Kolleg GmbH & Co. KG - Überörtliche Gemeinschaftspraxis Dres. Verpoort, Wierecky, Zeller, Hamburg

IPD SHARING:
Plan to Share IPD: Undecided